CLINICAL TRIAL: NCT06402500
Title: The Color Masking Potentials of a Bioactive Glass Adhesive and the Resin ICON on the White Spot Lesions. A Comparative Clinical Trial
Brief Title: Color Masking Potential of Bioactive and ICON Materials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JUST
Record Dates: First submitted 2024-04-15; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: White Spot Lesion of Tooth
Keywords: Resin infiltration; Incipient lesion; bioactive material; ICON infiltration resin
MeSH Terms: interventions — icon infiltrant

STUDY DESIGN:
Intervention Model Description: Split mouth study design, patients will be assigned to two different treatment protocols.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients who participated in the study and the assessor of the treatment outcome did not know the type of treatment procedure received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICON resin group (Experimental): Clean the white spot with prophylactic paste and then infiltrate the lesion with ICON resin.
  Interventions: Drug: Icon Infiltrant
- Bioactive resin group (Experimental): Clean the white spot with prophylactic paste and then infiltrate the lesion with bioactive resin.
  Interventions: Drug: Bioactive infiltrant

INTERVENTIONS:
Drug: Icon Infiltrant — White spot lesions are treated with the resin ICON (DMG, NJ, US) for masking their color. The mineral content will be measured in the lesion at baseline and after one month Quantitative light-induced fluorescence QLF.
  Other Names: ICON (DMG, NJ, US)
  Arms: ICON resin group
Drug: Bioactive infiltrant — White spot lesions are treated with HI-Bond universal bioactive resin (MEDICLUS, south Korea) for masking their color. Mineral content will be measured in the lesion at baseline and after one month Quantitative light-induced fluorescence QLF.
  Other Names: MEDICLUS, Cheongju-si, south Korea
  Arms: Bioactive resin group

SUMMARY:
The non cavitated white-spot lesion (WSL) occurs after sometime during fixed orthodontic treatments, and their treatment is mandatory before going into frank cavitation. The resin infiltration material (ICON, DMG, America) is considered to be the gold standard resin infiltrationmaterial used for WSL treatment. It is an efficient material in arresting WSLs and has high favorable esthetic recovery. Furthermore, biomaterials like bioactive glass adhesives HI-bond universal adhesive have always been used for replacement, repair and generation of dental hard tissues. The hypotheses of this study are:

1. There will be no differences in color masking effect on WSLs managed by bioactive glass adhesive or ICON resin infiltration.
2. There will be no significant addition of mineral content into WSLs after treating it with bioactive glass adhesive HI-Bond universal or with ICON.

DETAILED DESCRIPTION:
After sample size calculations were carried out a total sample size of 150 teeth will be included (75 teeth will be treated with ICON; and 75 other teeth will be treated with HI-Bond universal].

Split mouth study design involves treating WSLs in two different quadrants in each participant. Treatments will be done according to manufacturer's instruction. The WSLs in the teeth of one quadrant will receive treatments with the ICON (DMG, America) , and the others in the opposite quadrant will receive treatments with the bioactive glass adhesive HI-Bond universal (MEDICLUS, south Korea).

Before receiving the treatment, the WSLs will be tested at baseline by Quantitative light-induced fluorescence (QLF) device then the test will be repeated at 1-month after the treatment for the quadrant that received bioactive glass adhesive.

ELIGIBILITY:
Inclusion Criteria: Patients with teeth and WSL fullfiling the following criteria will be included in the study:

1. Anterior and premolar maxillary and mandibular teeth.
2. Teeth with no previous restorations.
3. post-orthodontic white spot lesions WSL with no adjacent restorations in the same tooth.
4. WSL on Labial surfaces of maxillary or mandibular anterior and premolars teeth.

Exclusion Criteria: The following will be excluded from the study,

1. Cavitated enamel surface that requires direct composite restorations.
2. Presence of developmental enamel defects on the proposed teeth.
3. Diabetic patients and patients with metabolic syndrome.
4. Pregnant ladies.
5. Smoker patients.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Color masking potential of ICON material in white spot lesions in permanent teeth. | 6 months
  Photographs will be taken before, immediately after treatment, and 1-month after treatment. These photographs will be used for evaluating of the esthetic outcome by two groups of subjects. The first group comprises the patients themselves. The second group includes dentists. Participants in the evaluation process will will be based on a 100-mm visual analogue scale (VAS). Participants will draw a line on the scale indicating their satisfaction. A line drawn between 0 - 5 cm will mean unsatisfactory outcome while that drawn between 5 - 10 cm will indicate satisfactory outcome.
Color masking potential of HI-Bond universal material in white spot lesions in permanent teeth. | 6 months
  Photographs will be taken before, immediately after treatment, and 1-month after treatment. These photographs will be used for evaluating of the esthetic outcome by two groups of subjects. The first group comprises the patients themselves. The second group includes dentists. Participants in the evaluation process will will be based on a 10-cm visual analogue scale (VAS). Participants will draw a line on the scale indicating their satisfaction. A line drawn between 0 - 5 cm will mean unsatisfactory outcome while that drawn between 5 - 10 cm will indicate satisfactory outcome.

SECONDARY OUTCOMES:
The remineralisation potential of HI-Bond universal material of white spot lesion (WSL) in permanent teeth. | 3 months
  Before receiving the HI-Bond material treatment, the WSL area will be measured by (QLF) device. The fluorescence intensities in the surrounding healthy enamel (baseline); and that in the white spot lesion are computed. The fluorescence loss is the difference of fluorescence intensities between the fluorescence of healthy enamel and that of the WSL.
  The same procedure and calculations are repeated after one month of treating the WSL with HI-Bond universal material.
  The fluorescence loss (ΔF) is typically reported as percentage (%) of fluorescence loss of that of the surrouding healthy enamel (baseline).
The remineralisation potential of HI-Bond universal material in the deepest point of the white spot lesion (WSL) in permanent teeth. | 3 months
  Before receiving the HI-Bond material treatment, the WSL area will be measured by (QLF) device. Then, the QLF software identifies and quantifies the fluorescence intensity at the area of most significant demineralization within the lesion which is marked by the maximum fluorescence loss within the lesion when compared to that of the surrounding health enamel.
  Deepest point in the lesion represents the maximum depth of fluorescence loss within the white spot lesion and is designated the symbol (ΔFMax).
  The ΔFMax represents the point within the white spot lesion where the demineralization is most severe, indicating the deepest point of mineral loss.
  The same procedure and calculations are repeated after one month of treating the WSL with HI-Bond universal material.
  Deepest point in the lesion (ΔFMax) is reported as a percentage (%) of fluorescence loss of that of surrounding healthy enamel (baseline).
The remineralisation potential of HI-Bond universal material on lesion area (pixels) of white spot (WSL) in permanent teeth. | 3 months
  Before receiving the HI-Bond material treatment, the Lesion area of the WSL is manually selected using (QLF) device. Then, the software identifies pixels with reduced fluorescence intensity compared to that of healthy surrounding enamel.
  The Lesion area (AΔF) is calculated by summing the total number of demineralized pixels identified within the white spot lesion region. Each pixel represents a unit of area. The area is generally expressed in pixels² (px²) by the software associated with QLF device.
  Through the software calibration this value can be converted into mm². The test will be repeated after 1-month of treatment with bioactive glass adhesive.
  When reporting the Lesion area (AΔF) in the context of QLF analysis, the unit is in pixels squared (px²).

CONTACTS AND LOCATIONS:
Overall Officials: Zakereyya SM Albashaireh, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan